CLINICAL TRIAL: NCT06620094
Title: The EFFECT of MOBILE APPLICATION USE on DIABETES CONTROL in DIABETIC PATIENTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Fidan Balkaya, Research Asistant, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Faculty of Nursing; TSA-2021-2582 (Other Grant/Funding Number: Inonu University of Scientific Research Project)
Record Dates: First submitted 2024-09-24; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Diabetes
Keywords: Diabetes mellitus, glycated hemoglobin A, mobile applications
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: This study is a pre-test, post-test randomized controlled experimental study. Therefore this study there is two groups: Intervention and control.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): This group, used mobile application and underwent routine controls.
  Interventions: Other: diabetes education videos
- Control Group (No Intervention): This group, underwent only routine controls.

INTERVENTIONS:
Other: diabetes education videos — In the initial meeting during the preparation phase, participants in the experimental group were informed about the notifications and diabetes education videos that would be sent to their phones. Afterward, the patients received three notifications daily, every day of the week. The first notification requested them to ;measure and record their fasting and postprandial blood sugar in the morning; The second notification instructed them to ;exercise for at least 30 minutes a day.; The third notification asked them to ;record the foods they consumed and their quantities, and to measure and record their evening fasting and postprandial blood sugar, as well as their blood sugar before going to bed.; Additionally, during their routine outpatient follow-ups, the results of their tests (A1C, BMI, total cholesterol, HDL, LDL, triglycerides), blood pressure, and weight measurements were recorded. Furthermore, three times a week, participants were asked to ;measure and record their blood pressur
  Arms: Intervention Group

SUMMARY:
Objective:This study aims to determine the effect of a mobile application on diabetes control in patients with Type 2 diabetes.

Methods:This study is a randomized controlled trial with a pre-test and post-test design. The study population consists of Type 2 diabetes patients who applied to the Endocrinology Clinic of Malatya Turgut Özal Medical Center. A total of 70 participants were included in the study. Data were collected face-to-face using a demographic data collection form, a diabetes diagnosis and follow-up form, and the Turkish Multidimensional Diabetes Scale. The data were analyzed using paired t-tests and independent samples t-tests to compare means, counts, and percentages in dependent and independent groups.

DETAILED DESCRIPTION:
Type of Study: This study is a pre-test, post-test randomized controlled experimental study.

Population and Sample of the Study: The population of the study consisted of individuals with type 2 diabetes who applied to the Endocrinology Clinic of Malatya Inonu University Turgut Ozal Medical Center between May 2021 and December 2021. The sample included patients who met the inclusion criteria during the dates of the study and who applied to the Endocrinology Clinic. The power analysis used to determine the sample size was calculated with a 5% margin of error, 95% confidence interval at a two-sided significance level, and 80% population representation capacity, with 50 diabetic individuals for each group (50 experimental, 50 control). However, the study was completed with 38 individuals in the experimental group and 32 in the control group.

Inclusion Criteria:

Having been diagnosed with type 2 diabetes mellitus for at least 6 months. Being between the ages of 40-65. Receiving oral antidiabetic treatment. Having an A1C value between 7%-10%. Owning a mobile phone capable of receiving and playing video messages. Not having sensory impairments, such as hearing or speech loss, or psychiatric problems that prevent communication.

Exclusion Criteria:

Inability to use the mobile application. Patients with a psychological diagnosis according to records. Patients using insulin. Having an A1C value above 10%. Having an infection requiring medication. Randomization: Care was taken to ensure that the two groups were homogeneous by considering all variables. The assignment of diabetic patients to the experimental and control groups was done through randomization to avoid bias. The randomization was carried out using the Random Integer Generator method in the Numbers section of the random.org website, where columns with five groups between 1-100 were generated. Patients who applied to the Endocrinology Clinic were randomized to numbers 1 and 2, based on which they were assigned to the groups. The determination of which number corresponded to the experimental or control group was made by drawing lots at the beginning of the study.

Data Collection Tools: Two data collection tools were used to collect the data.

Diabetes Patient Identification and Monitoring Form: This form, prepared by the researchers with the help of literature reviews and expert opinions, consists of three parts. The first part contains 11 items used to determine the socio-demographic characteristics of the patient. The second part consists of 32 items that question the patient's diabetes-related characteristics, such as diabetes type, treatment method, complications, treatment follow-up routines, nutrition, exercise routines, foot care, diabetes-related knowledge, and habits. The third part consists of 9 items that question the metabolic control characteristics of diabetic individuals, such as fasting blood sugar, A1C, total cholesterol, LDL, HDL, triglycerides, blood pressure, height, weight, and body mass index.

Turkish Multidimensional Diabetes Questionnaire (T-MDQ): This scale was developed by Talbot and colleagues in 1997. The Turkish validity and reliability of the scale were conducted by Coşansu and Erdoğan in 2010. The scale consists of 40 items, 7 sub-dimensions, and 3 sections. The scale has no total score, and each sub-dimension is evaluated separately.

Section: Focuses on the general perception of diabetes and social support. This section consists of three sub-dimensions and 16 items. The Perceived Barrier sub-dimension consists of 9 items questioning how much the patient's daily activities such as work, social, and leisure activities are negatively affected and limited due to diabetes. The Perceived Severity consists of 3 items measuring the degree of the patient's perception of the seriousness of diabetes. The Perceived Social Support sub-dimension consists of 4 items questioning the patient's perceived social support from important people in their life, such as family, friends, and healthcare professionals. In the first section, responses are obtained with a 7-point Likert scale (0-none, 6-very much). The scores of the items answered by the individual for each sub-dimension are summed and divided by the number of items answered to obtain an average score. Higher scores indicate higher perceived barriers, social support, and severity levels.

Section: Investigates the behaviors of the patient's spouse or someone significant to them that either support or fail to support the patient's self-care activities for diabetes. This section consists of two sub-dimensions and 12 items. Positive Supportive Behaviors consist of 8 items aimed at identifying positive behaviors of the patient's spouse or significant other that support the patient's management of diabetes. The Misleading Supportive Behaviors sub-dimension consists of 4 items aimed at identifying supportive but bothersome and unhelpful behaviors of the patient's spouse or significant other. Responses in the second section are recorded on a 7-point Likert scale (0-never, 6-always). Individuals living alone do not fill out this section.

Section: Measures the individual's perception of self-efficacy and outcome expectations related to disease management. This section consists of two sub-dimensions and 13 items. The Perceived Self-Efficacy sub-dimension consists of 7 items that determine the individual's confidence in performing self-care activities for their illness. Responses are recorded on a Likert scale (0-not confident at all, 100-very confident). The Perceived Outcome Expectation sub-dimension consists of 6 items that evaluate the individual's perception of the effectiveness of self-care behaviors and treatment in achieving metabolic control and preventing complications. Responses are recorded on a Likert scale (0-not important at all, 100-very important). Higher scores indicate higher perceived self-efficacy and outcome expectations.

Data Collection: The data of the study were collected through face-to-face interviews by the researcher with type 2 diabetic patients who applied to the Endocrinology Clinic between May 2021 and December 2021. Patients meeting the inclusion criteria were included in the study.

Initially, data collection forms (survey form and T-MDQ) were applied to the patients in the experimental and control groups. Additionally, patients' test results (A1C, glucose, total cholesterol, HDL, LDL, triglycerides), blood pressure, height, and weight measurements were recorded during routine outpatient follow-ups. The experimental group received education and follow-up for three months through a mobile application prepared for diabetic patients. At the end of this period, the T-MDQ, routine test results (A1C, glucose, total cholesterol, HDL, LDL, triglycerides), blood pressure, height, and weight measurements were applied again to both the experimental and control groups.

Intervention: During the initial interview with the experimental group, participants were informed about notifications and diabetes education videos that would be sent to their phones. Following this, notifications were sent three times a day, every day of the week. The first notification asked the patient to ;measure and record their fasting and postprandial blood sugar in the morning," the second instructed to "exercise for at least 30 minutes a day," and the third asked them to "record the foods and amounts they ate, measure and record their evening fasting and postprandial blood sugar, and measure and record their blood sugar before going to bed." The results of their routine outpatient tests (A1C, BMI, total cholesterol, HDL, LDL, triglycerides), blood pressure, and weight measurements were recorded. In addition, three times a week, participants were asked to "measure and record their blood pressure and weight, and log the recorded information in the app each time; During the three-month period, individuals continued their routine outpatient follow-ups.

Control Group: During the first meeting, after being informed about the study, data collection forms (survey form and Turkish Multidimensional Diabetes Questionnaire) were applied to the control group. The results of the routine outpatient tests (A1C, glucose, total cholesterol, HDL, LDL, triglycerides) were recorded. Blood pressure, height, and weight measurements were taken, and the first interview was completed. The control group continued their routine outpatient follow-ups. During the second meeting, which took place three months later, the data collection forms were applied again. The results of routine outpatient tests (A1C, BMI, total cholesterol, HDL, LDL, triglycerides) were written down, and blood pressure and weight measurements were taken and recorded.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with type 2 diabetes mellitus for at least 6 months. Being between the ages of 40-65. Receiving oral antidiabetic treatment. Having an A1C value between 7%-10%. Owning a mobile phone capable of receiving and playing video messages. Not having sensory impairments, such as hearing or speech loss, or psychiatric problems that prevent communication.

Exclusion Criteria:

* Inability to use the mobile application. Patients with a psychological diagnosis according to records. Patients using insulin. Having an A1C value above 10%. Having an infection requiring medication.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-05-30 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
A1C levels | up to seven months
  Hemoglobin A1C (HbA1C): HbA1C is a blood test that measures the average blood glucose levels over the past two to three months by determining the percentage of glycated hemoglobin in the blood. It is commonly used to diagnose diabetes and assess the effectiveness of diabetes management. An HbA1C level below 5.7% is considered normal, between 5.7% and 6.4% indicates prediabetes, and a level of 6.5% or higher indicates diabetes.

CONTACTS AND LOCATIONS:
Overall Officials: Rukuye AYLAZ, Prof. Dr., Study Director — Inonu University Faculty of Nursing
Locations (1):
- Inonu University, Malatya, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data are not open to public due to confidentiality and ethical restrictions.